CLINICAL TRIAL: NCT04014660
Title: Prevention av Autoimmunitet Med Laktobaciller (in English; Prevention of Autoimmunity With Lactobacilli)
Brief Title: Prevention av Autoimmunitet Med Laktobaciller
Acronym: PAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-02322
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Celiac Disease in Children; Type 1 Diabetes; Thyroid
Keywords: celiac disease autoimmunity; islet autoimmunity; auto-antibodies
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Thyroid Diseases | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): The participants in this group are provided with a dietary supplement (capsules) containing freeze dried bacteria (active lactobacilli culture) mixed with corn starch, for daily intake (1 capsule per day).
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): The participants in this group are provided with a dietary supplement (capsules) containing corn starch only, for daily intake (1 capsule per day).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The probiotic product consists of two different bacterial strains, L.plantarum Heal 9 and L.paracasei 8700:2
  Arms: Probiotic group
Dietary Supplement: Placebo — The placebo supplement consists of corn starch only.
  Arms: Placebo group

SUMMARY:
The incidence of autoimmune diseases (celiac disease, type 1 diabetes, thyroid disease) have increased over the past 30 years. Although most autoimmune diseases have a strong link to different risk genes, the rapid increase is thought to be due to changes in environmental factors. There is currently no cure for autoimmune diseases, but the treatment is lifelong and either involves suppressing the inflammation and / or substituting the organs that are affected to maintain vital functions. Being able to predict who is affected and identifying factors that trigger autoimmunity is necessary for developing new treatment methods that prevent the occurrence of autoimmune diseases. The bacterial flora's composition in the gut can affect both the intestinal barrier properties and the immune system's response to various dietary components. An adverse composition of the intestinal flora can activate parts of the immune system that are involved in chronic inflammation in celiac disease and inflammatory bowel disease. Probiotics are defined as living microorganisms which, when ingested in sufficient amounts, produce a health effect (FAO / WHO). The aim of the study is to investigate whether a daily oral intake of a mixture of L.paracasei and L.plantarum can affect the autoimmune process in children who are screened positive for any of the autoantibodies associated with development of celiac disease, type 1 diabetes and / or thyroid disease. Our hypothesis is that lactobacilli can directly regulate the autoimmune process in the small intestinal mucosa by stimulating regulatory T-cells, but also by affecting the permeability of the small intestinal mucosa by of antigen that stimulates specific T-cells.

DETAILED DESCRIPTION:
The incidence of autoimmune diseases (celiac disease, type 1 diabetes, thyroid disease) have increased over the past 30 years. Although most autoimmune diseases have a strong link to different risk genes, the rapid increase is thought to be due to changes in environmental factors. There is currently no cure for autoimmune diseases, but the treatment is lifelong and either involves suppressing the inflammation and / or substituting the organs that are affected to maintain vital functions. Being able to predict who is affected and identifying factors that trigger autoimmunity is necessary for developing new treatment methods that prevent the occurrence of autoimmune diseases.

The bacterial flora's composition in the gut can affect both the intestinal barrier properties and the immune system's response to various dietary components. An adverse composition of the intestinal flora can activate parts of the immune system that are involved in chronic inflammation in celiac disease and inflammatory bowel disease.

Probiotics are defined as living microorganisms which, when ingested in sufficient amounts, produce a health effect (FAO / WHO). Certain probiotic strains has been used to hamper pro-inflammatory immune system triggered by gluten protein in conjunction with celiac disease. Earlier studies have shown that Lactobacillus reduced the permeability in the small intestinal mucosa. But to our knowledge, no randomized clinical trials have tested the effect on probiotic supplementation and development of autoimmune disease such as celiac disease.

The aim of the study is to investigate whether a daily oral intake of a mixture of L.paracasei and L.plantarum can affect the autoimmune process in children who are screened positive for any of the autoantibodies associated with development of celiac disease, type 1 diabetes and / or thyroid disease. Our hypothesis is that lactobacilli can directly regulate the autoimmune process in the small intestinal mucosa by stimulating regulatory T-cells, but also by affecting the permeability of the small intestinal mucosa by of antigen that stimulates specific T-cells.

The aims of this study are:

* will supplementation of L.paracasei and L.plantarum during a 12 month period compared to placebo increase the levels of regulatory T-cells (CD4+CD25+) and decrease B-cells and/or NK-cells in children and adolescents screened persistent positive with auto-antibodies associated with celiac disease, type 1 diabetes and / or thyroid disease?
* will supplementation of L.paracasei and L.plantarum during a 12 month period compared to placebo increase the abundance of bacteroides in gut and oral cavity in children and adolescents screened persistent positive with auto-antibodies associated with celiac disease, type 1 diabetes and / or thyroid disease?
* will supplementation of L.paracasei and L.plantarum during a 12 month period compared to placebo lower the levels of auto-antibodies associated with celiac disease, type 1 diabetes and / or thyroid disease in children and adolescents with persistent positive auto-antibodies.

A total of 200 children genetically at-risk for celiac disease, type 1 diabetes and thyroid disease who are persistent positive for any of the following auto-antibodies will be invited to the study.

Participants who signed a informed consent will be randomized (double blinded) into the probiotic or placebo group. A venous blood sample, saliva- and feces sample will be collected at every clinic visit, 3 months apart (0, 3, 6, 9 and 12 months). A short questionnaire collecting information about illnesses, medication- and dietary supplement use, food habits, and demographic factors will be used.

Blood sample will be analyzed for auto-antibodies (tTGA, GADA, IA-2A, IAA, Zn-T8A, and TPOA). FACS analyses will be used for a panel of inflammatory markers (CD3, CD4, CD8, CD25 etc). Feces- and saliva samples will be analysed using T-RFLP (PCR) of 16S rRNA.

The benefit if this study are the increased knowledge about specific probiotics strains impact on autoimmunity in genetically at-risk children, and hopes of reducing the risk for developing autoimmune diseases as celiac disease, type 1 diabetes and thyroid disease.

ELIGIBILITY:
Inclusion Criteria:

* Screened persistent positive for any of the auto-antibodies associated with celiac disease (tTGa), type 1 diabetes (IAA, GADA, IA-2A, Zn-T8) and/or thyroid disease (TPOA)

Exclusion Criteria:

* None

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 202 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Autoimmunity | 12 months
  To study levels of auto-antibodies (tTGA, GADA, IA-2, IAA, ZnT8a, TPOA) genetically at-risk children. (Blood sample will be analyzed for auto-antibodies (tTGA, GADA, IA-2A, IAA, Zn-T8A, and TPOA)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Agardh, PhD, Principal Investigator — Dep Clinical Sciences, Lund University
Locations (1):
- Clinical Research Center (CRC), Bldng 60:11, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eun CS, Kim YS, Han DS, Choi JH, Lee AR, Park YK. Lactobacillus casei prevents impaired barrier function in intestinal epithelial cells. APMIS. 2011 Jan;119(1):49-56. doi: 10.1111/j.1600-0463.2010.02691.x. Epub 2010 Oct 25. PMID 21143526
- [Result] Falk A, Olsson C, Ahrne S, Molin G, Adawi D, Jeppsson B. Ileal pelvic pouch microbiota from two former ulcerative colitis patients, analysed by DNA-based methods, were unstable over time and showed the presence of Clostridium perfringens. Scand J Gastroenterol. 2007 Aug;42(8):973-85. doi: 10.1080/00365520701204238. PMID 17613928
- [Result] Laparra JM, Sanz Y. Bifidobacteria inhibit the inflammatory response induced by gliadins in intestinal epithelial cells via modifications of toxic peptide generation during digestion. J Cell Biochem. 2010 Mar 1;109(4):801-7. doi: 10.1002/jcb.22459. PMID 20052669
- [Result] Lavasani S, Dzhambazov B, Nouri M, Fak F, Buske S, Molin G, Thorlacius H, Alenfall J, Jeppsson B, Westrom B. A novel probiotic mixture exerts a therapeutic effect on experimental autoimmune encephalomyelitis mediated by IL-10 producing regulatory T cells. PLoS One. 2010 Feb 2;5(2):e9009. doi: 10.1371/journal.pone.0009009. PMID 20126401
- [Result] Llopis M, Antolin M, Carol M, Borruel N, Casellas F, Martinez C, Espin-Basany E, Guarner F, Malagelada JR. Lactobacillus casei downregulates commensals' inflammatory signals in Crohn's disease mucosa. Inflamm Bowel Dis. 2009 Feb;15(2):275-83. doi: 10.1002/ibd.20736. PMID 18839424
- [Result] Wang M, Ahrne S, Antonsson M, Molin G. T-RFLP combined with principal component analysis and 16S rRNA gene sequencing: an effective strategy for comparison of fecal microbiota in infants of different ages. J Microbiol Methods. 2004 Oct;59(1):53-69. doi: 10.1016/j.mimet.2004.06.002. PMID 15325753
- [Result] Wang M, Ahrne S, Jeppsson B, Molin G. Comparison of bacterial diversity along the human intestinal tract by direct cloning and sequencing of 16S rRNA genes. FEMS Microbiol Ecol. 2005 Oct 1;54(2):219-31. doi: 10.1016/j.femsec.2005.03.012. PMID 16332321